CLINICAL TRIAL: NCT01794273
Title: Compared Efficacy and Tolerance of Two Vasopressors Used to Treat Preoperative Hypotension During Carotid Surgery. Prospective Randomised Controlled and Single Centre Trial
Brief Title: Compared Efficacy and Tolerance of Two Vasopressors Used to Treat Preoperative Hypotension During Carotid Surgery
Acronym: VP-hTA-XCar
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CHU-0147; 2012-001827-11
Record Dates: First submitted 2013-02-15; First posted 2013-02-18 (Estimated); Last update posted 2018-09-24 (Actual); Status verified 2018-09

CONDITIONS: Endovascular Carotid Surgery; Preoperative Hypotension
Keywords: Ephedrine; Phenylephrine; Vasopressor; Carotid surgery; Hypotension; Haemodynamics; Brain ischemia; Tissue perfusion; Stroke; anaesthesia
MeSH Terms: conditions — Hypotension; Brain Ischemia; Stroke | interventions — Ephedrine; Phenylephrine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- ephedrine (Experimental): This is a randomised trial comparing ephedrine and phenylephrine as used for accidental hypotension occurring during carotid surgery, on cerebral perfusion, assessed by near-infrared spectroscopy (NIRS).
  Interventions: Drug: ephedrine and phenylephrine
- phenylephrine (Experimental): This is a randomised trial comparing ephedrine and phenylephrine as used for accidental hypotension occurring during carotid surgery, on cerebral perfusion, assessed by near-infrared spectroscopy (NIRS).
  Interventions: Drug: ephedrine and phenylephrine

INTERVENTIONS:
Drug: ephedrine and phenylephrine

SUMMARY:
The effects on brain perfusion of the two currently vasopressors used to treat accidental hypotension occurring during carotid surgery (i.e. ephedrine and phenylephrine) is not known, but a disadvantage to use phenylephrine is suspected, due to its mechanism of action and according to published reports

DETAILED DESCRIPTION:
This is a randomised trial comparing ephedrine and phenylephrine as used for accidental hypotension occurring during carotid surgery, on cerebral perfusion, assessed by near-infrared spectroscopy (NIRS).

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 ASA score I-III Planned carotid endarteriectomy under general anaesthesia Hypotension defined as SAP < 90 mm Hg during general anaesthesia Informed consent to the trial Protected by the French health welfare

Exclusion Criteria:

* Emergency surgery Cardiac arrythmia Pregnancy or breastfeeding Allergy to the tested treatment Allergy to hydroxyethylstarch Allergy to the glue of the NIRS's electrodes Current medication: MAOI, intranasal vasopressors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2013-07 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Cerebral oxygen saturation (SctO2) | at day 1

SECONDARY OUTCOMES:
Incidence of post-treatment hypotension | At day 1
Incidence of post-treatment bradycardia | at day 1
Postoperative morbidity: cardiovascular, cerebral, renal, surgical | at day 1
Postoperative recovery | at day 1

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte BAUD, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Background] Aliane J, Duale C, Guesmi N, Baud C, Rosset E, Pereira B, Bouvier D, Schoeffler P. Compared effects on cerebral oxygenation of ephedrine vs phenylephrine to treat hypotension during carotid endarterectomy. Clin Exp Pharmacol Physiol. 2017 Jul;44(7):739-748. doi: 10.1111/1440-1681.12759. PMID 28378467